CLINICAL TRIAL: NCT02839603
Title: Asymptomatic Leishmania Infection and Burden of Visceral Leishmaniasis in HIV-infected Individuals in North West Ethiopia: a Pilot Study
Brief Title: Asymptomatic Leishmania Infection in HIV Patients
Status: Terminated | Type: Observational
Why Stopped: Aim to assess feasibility achieved, larger project starting earlier than anticipated
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University of Gondar (Other); Addis Ababa University (Other); Metema District Hospital, Metema, Ethiopia (Unknown)
Responsible Party: Sponsor
Other Study IDs: 920/13
Record Dates: First submitted 2016-07-12; First posted 2016-07-21 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Visceral Leishmaniasis
Keywords: Visceral leishmaniasis; HIV co-infection; Asymptomatic
MeSH Terms: conditions — Leishmaniasis, Visceral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Plasma Whole blood Urine Stool
Oversight: Data Monitoring Committee: No

SUMMARY:
To collect pilot data on the prevalence and incidence of asymptomatic Leishmania donovani infection in HIV infected individuals in a visceral leishmaniasis (VL)-HIV endemic region to inform the feasibility of a larger study exploring a screen and treat strategy for VL in HIV co-infected individuals in East-Africa (Ethiopia).

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* without a history of VL in the last 5 years
* stable residents of a VL-endemic area
* willing to participate and giving free informed consent

Exclusion Criteria:

* younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult individuals enrolled in HIV care in Metema hospital
Sampling Method: Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
The proportion of individuals with L.donovani asymptomatic infection at baseline in HIV coinfected adults enrolled in HIV care in a VL-HIV endemic region in North-West Ethiopia. | End of study (2 years)
  Proportion of individuals with asymptomatic infection, defined as positivity on any of the leishmanial markers (PCR, urine antigen or serology)

SECONDARY OUTCOMES:
The proportion of individuals with asymptomatic infection during follow-up in HIV coinfected adults enrolled in HIV care in a VL-HIV endemic region in North-West Ethiopia | End of study (2 years)
  Proportion of individuals with asymptomatic infection during follow-up, defined as positivity on any of the leishmanial markers (PCR, urine antigen or serology) amongst those without asymptomatic infection during the cross-sectional evaluation.
Proportions of individuals with a positive test on a specific leishmanial marker to describe the pattern of asymptomatic infection. | End of study (2 years)
Proportion of asymptomatic infected patients in clinical determinant groups. | End of study (2 years)
  Clinical determinant groups are constructed with key clinical characteristics and history
Total proportion of baseline asymptomatic infected patients, with positive infection status at 3, 6, 9 and 12 months follow-up. | 3, 6, 9 and 12 months of follow-up
Proportion of baseline asymptomatic infected patients, with positive infection status for each baseline leishmanial marker at 3, 6, 9 and 12 months | 3, 6, 9 and 12 months of follow-up
Proportion of individuals developing VL within the following year (= One-year risk of VL) | End of study (2 years)
  VL will be diagnosed as per national guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Metema District Hospital, Metemma, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Griensven J, van Henten S, Mengesha B, Kassa M, Adem E, Endris Seid M, Abdellati S, Asefa W, Simegn T, Debasu D, Bogale T, Gedamu Y, Van Den Bossche D, Adriaensen W, Van der Auwera G, Cnops L, Vogt F, Diro E. Longitudinal evaluation of asymptomatic Leishmania infection in HIV-infected individuals in North-West Ethiopia: A pilot study. PLoS Negl Trop Dis. 2019 Oct 8;13(10):e0007765. doi: 10.1371/journal.pntd.0007765. eCollection 2019 Oct. PMID 31593563